CLINICAL TRIAL: NCT03570112
Title: Evaluation of the Natural History and Vertical Transmission of Chronic Hepatitis C Virus Infection in Pregnancy With Targeted Elimination by Postpartum Treatment
Brief Title: Transmission of Chronic Hepatitis C in Pregnancy
Status: Completed | Type: Observational
Sponsor: The Christ Hospital (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, John Cafardi, Dr. John Cafradi, MD, Infectious Disease Specialist, The Christ Hospital
Other Study IDs: 18-08
Record Dates: First submitted 2018-06-06; First posted 2018-06-26 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C; Pregnancy Complications; Vertical Disease Transmission
MeSH Terms: conditions — Hepatitis C; Pregnancy Complications | interventions — velpatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant Women with Hep C: SOF/VEL Therapy-sofosbuvir 400mg, velpatasvir 100mg, once daily for 12 weeks at 24 weeks post partum
  Interventions: Drug: SOF/VEL- sofosbuvir 400mg and velpatasvir 100mg

INTERVENTIONS:
Drug: SOF/VEL- sofosbuvir 400mg and velpatasvir 100mg — sofosbuvir 400mg and velpatasvir 100mg once daily for 12 weeks
  Other Names: Epclusa

SUMMARY:
This is a multicenter, non-comparative, observational study that will recruit women with singleton pregnancy and chronic HCV infection to determine the natural history of chronic HCV in pregnancy and the rate of vertical transmission to their infants. All participants will be offered curative therapy with sofosbuvir/velpatasvir (Epclusa ®) after delivery and the cessation of breastfeeding. Subjects may be enrolled at any time after conception up through 36 weeks gestation. The management of subjects in pregnancy will be in accordance with ACOG guidelines and individual clinical judgment, however testing will include, but not be limited to, testing for HCV infection, HIV infection, HBV infection, HSV infection, group B Streptococcal colonization, HCV genotype, HCV viral load, as well as assessment of hepatic and renal function. Subjects will be followed on a schedule that is determined by their obstetric care providers throughout their pregnancy. Following delivery, infants will be evaluated at 12, 24 and 48 weeks of age, with testing for HCV RNA to be obtained at each evaluation. Vertical transmission is defined as two positive HCV RNA PCR tests, at least one before the 48 week infant visit, and again at the 12-month follow-up infant visit.

DETAILED DESCRIPTION:
The treatment of chronic hepatitis C virus infection has dramatically advanced in recent years, with the availability of multiple interferon-free treatment regimens that result in cure in over 95% of treatment naïve individuals with 8 -12 weeks of therapy. Despite these advances, however, the natural history and treatment of HCV remains undefined in several populations, including pregnancy. In particular, rates of vertical (mother to child) transmission, perinatal and neonatal morbidity, assessment of disease severity (fibrosis) in pregnancy and timing of treatment are not well understood.

At least 2.3 million people in the United States and 185 million people worldwide are believed to have chronic HCV infection, although as it is frequently asymptomatic until the development of end-stage liver disease (ESLD), this may be a significant underestimate. Between 2012 and 2014 the HCV detection rate among women of childbearing age increased by 22% nationally and over 200% in Kentucky, while the proportion of children born to HCV infected women increased 68% nationally and 128% in Kentucky.

Currently, in the United States, the overall rate of children born to HCV infected women is 3.4 per 1,000 live births, with the highest rate in West Virginia, with 22.4 per 1,000 live births occurring to HCV-infected women. Overall, the number of HCV infected reproductive age women has doubled from 2006 to 2014, with an estimated 29,000 HCV infected women giving birth and 1,700 infants vertically infected each year, according to previous estimates of vertical transmission.The true incidence of vertical transmission of HCV is unknown, although the most commonly cited meta-analysis reported a mean transmission rate of 5.8% in HIV-negative women and 10.8% in HIV-positive women.

The timing of vertical transmission is also not well characterized. There is limited data regarding the course of chronic hepatitis C during pregnancy, HCV viral loads appear to peak during third trimester. Both utero and peripartum transmission appear possible, while breastfeeding does not appear to be a risk factor. It appears that between 80 and 90% of children who acquire hepatitis C via vertical transmission will develop chronic infection. However, as sequelae of infection are not commonly observed in childhood, and appropriate testing of exposed children is poor, this may not be a true reflection of actual prevalence.

The current AASLD/IDSA HCV Guidelines recommend all children born to HCV infected women be tested, but they do not specify when or in what manner.

Maternal HCV infection has been shown to contribute to worsened perinatal and neonatal outcomes in the absence of vertical transmission. It is associated with increased rates of intrauterine fetal death, preterm delivery, low birth rate, increased risk for adverse neonatal neurological outcomes, increased infant feeding difficulties and subsequent maternal infertility.

Although there is sufficient time between the end of the first trimester and delivery to provide curative therapy during pregnancy, no safety studies in pregnancy have been done. Therefore, this study will offer curative DAA therapy to HCV infected Moms with the fixed dose combination of sofosbuvir/velpatasvir (SOF/VEL) after the cessation of breastfeeding. This combination of sofosbuvir, a nucleotide inhibitor of the NS5B RNA-dependent RNA polymerase, and velpatasvir, an inhibitor of the NS5A transcriptional activator, is approved for the treatment of chronic HCV infection due to genotypes 1 through 6.

Given the gaps in the investigator's understanding of HCV vertical transmission rates, HCV-associated perinatal complications, and marked increases in both the number of women with chronic HCV infection giving birth and the number of children under two years old testing positive for HCV, this study will help to both better characterize the natural history of HCV in pregnancy and ultimately, to facilitate its elimination when women are screened for chronic HCV as part of routine gynecologic care and are offered curative therapy prior to conception (or as part of prenatal care and when dosing during pregnancy can be safely undertaken).

All participants will be offered curative therapy with sofosbuvir/velpatasvir (Epclusa ®) after delivery and the cessation of breastfeeding. Subjects may be enrolled at any time after conception up through 36 weeks gestation. The management of subjects in pregnancy will be in accordance with ACOG guidelines and individual clinical judgment, however testing will include, but not be limited to, testing for HCV infection, HIV infection, HBV infection, HSV infection, group B Streptococcal colonization, HCV genotype, HCV viral load, as well as assessment of hepatic and renal function. Staging of hepatic fibrosis must be performed within 12 months prior to initiation of SOF/VEL. Acceptable methods of staging include transient elastography or liver biopsy. If elastography is performed, it must be performed either prior to pregnancy or at least 12 weeks following delivery, due to pregnancy-related changes in hepatic stiffness. Subjects will be followed on a schedule that is determined by their obstetric care providers throughout their pregnancy. Data from clinical and laboratory records regarding the participants pregnancy and delivery, and their infant's medical record from the infant's pediatrician from birth to 12 months of age will be collected. Following delivery, infants will be evaluated at 12, 24 and 48 weeks of age, with testing for HCV RNA to be obtained at each evaluation. Vertical transmission is defined as two positive HCV RNA PCR tests, at least one before the 48 week visit, and again at the 12-month follow-up infant visit.At 24 weeks following delivery, participants will begin therapy with sofosbuvir/velpatasvir (SOF/VEL) once daily for 12 weeks. Therapy will not be initiated until cessation of breastfeeding. Participants will be evaluated at the initiation of SOF/VEL therapy, at 4 and 8 weeks after starting therapy, as well as 12 weeks following completion of therapy for determination of SVR-12. Quantitative measurement of HCV RNA will be obtained at each visit, as well as evaluation of renal and hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Chronic HCV infection, as defined by positive HCV antibody with confirmation of positive HCV RNA PCR at least 6 months apart, per 2017 AASLD/IDSA criteria. Infection with any genotype (including mixed genotypes) is permitted.

  * If the diagnosis of chronic HCV is not established by two positive viral load (RNA PCR) tests 6 months apart, subjects may be enrolled and followed until the 6-month test is performed. If the follow-up viral load test is negative (i.e. the woman had acute infection that has cleared), the participant will be excluded from further study participation. All participants excluded for this reason will be replaced.
* Singleton pregnancy, up to and including 36 weeks' gestation, as documented by fetal ultrasound at any time during the pregnancy.
* Willing and able to understand and sign the informed consent form
* Willing and able to sign release of Information forms for their own medical and obstetric care and for their infant's neonatal and pediatric care for one year following delivery, or when the last study viral load test is performed, whichever comes later.

Exclusion Criteria:

* Co-infection with chronic hepatitis B.
* Active injection drug use, defined as the parenteral use of any substance for non-medicinal purposes in the previous 60 days. Potential subjects who have a history of active injection drug use will be referred to both syringe services programs to prevent the acquisition of HIV and HBV and to substance abuse treatment. Potential subjects who have injected within the last 60 days may be re-screened if they participate in a drug treatment program, subject to the discretion of the investigator.
* Decompensated cirrhosis, as determined by clinical history or examination
* Any major medical comorbidity that may confound assessment, such as cardiomyopathy, pulmonary hypertension, type 1 diabetes mellitus or similar serious medical conditions at the discretion of the investigator. Gestational diabetes mellitus or co-infection with HIV are not criteria for exclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with singleton pregnancy and chronic HCV infection
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the rate of vertical transmission | 12 months of age
  Evaluate the rate of vertical transmission in infants born to HCV infected mothers by detection of HCV RNA in the infant prior to and again at 12 months of age.

SECONDARY OUTCOMES:
SVR12 | 12 weeks post treatment
  Evaluate SVR12 - Hepatitis C undetectable
Pre-Term Birth | 12 weeks post partum
  Defined as delivery between 20 and 37 weeks
Cholestasis of pregnancy | 12 weeks post partum
  Defined by the Society for Maternal Fetal Medicine, consisting of pruritis, absence of rash, serum bile acids > 10umol/liter with resolution following delivery
Low Birth Weight | 12 weeks of age
  Defined by the World Health Organization, infant weighing 2,499 grams or less at birth regardless of gestational age
Presence and severity of NAS/NOWS | 12 weeks of age
  Neonatal abstinence syndrome(NAS)/ neonatal opioid withdrawal syndrome(NOWS) by modified Finnegan Neonatal Abstinence Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: John Cafardi, MD, Principal Investigator — The Christ Hospital
Locations (1):
- Lindner Research Center at the Christ hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No